CLINICAL TRIAL: NCT03119909
Title: Cognitive Adaptation and Frontal Cortex
Brief Title: Cognitive Adaptation
Acronym: ADAPCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0683
Record Dates: First submitted 2017-03-09; First posted 2017-04-19 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: fMRI; cingulate cortex; adaptation; frontal cortex

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Learning of actions-events associations (Other): Each subject will conduct 4 sessions, i.e. a training session and three fMRI sessions. The first session will consist in training the subject to carry out the different behavioral tasks that he will then have to perform during the sessions of fMRI.
  Interventions: Other: First session of fMRI: localization of the premotor areas of the medial frontal cortex; Other: Second fMRI session; Other: Third fMRI Session; Other: Training fMRI session
- Learning of action-event associations not linked to action (Other): This study is divided into two parts: a pilot behavioral study to determine the learning characteristics of non-action events and an fMRI study to study the neural networks involved in this type of learning.
  30 subjects will participate in the behavioral study and 60 will participate in the fMRI study)
  Interventions: Other: Pilot behavioral study; Other: fMRI Study

INTERVENTIONS:
Other: First session of fMRI: localization of the premotor areas of the medial frontal cortex — Subjects should perform simple tasks to map the premotor areas of the medial frontal cortex. In this context, they will have to perform hand, tongue, ocular movements for about 20s. Additionally, as part of a control condition, they will need to perform eye fixation on a cross shown at the center of the screen for about 20s.
  Arms: Learning of actions-events associations
Other: Second fMRI session — The subjects will position their left and right thumbs on response buttons. Each trial will begin with the appearance of one of 2 possible indexes. It will be an unknown abstract visual stimulus). After a variable delay of 0.5 to 6s (average = 2s), a blue or yellow circle will appear on the left or right of the screen.
  Arms: Learning of actions-events associations
Other: Third fMRI Session — This session is identical to the second session but the subject will have to respond by performing saccadic ocular responses.
  Arms: Learning of actions-events associations
Other: Training fMRI session — The training session will consist in training the subject to carry out the different behavioral tasks that he will then have to perform during the sessions of fMRI.
  Arms: Learning of actions-events associations
Other: Pilot behavioral study — In a pilot study, 30 subjects will participate in a behavioral study (2 sessions of 2 hours each) aimed at establishing the learning characteristics of the different types of rare events unrelated to actions (visual and sensorimotors on the hand).
  Arms: Learning of action-event associations not linked to action
Other: fMRI Study — Each subject will participate in 2 fMRI sessions of about 2 hours each: a first session in which a first version of the task will be presented and a second session in which the second version of the task will be presented.
  Arms: Learning of action-event associations not linked to action

SUMMARY:
A hallmark of our survival in the real world and of our capacity to navigate the complex social interactions of human society is our ability to show behavioral adaptation. Adaptation can be necessary for a number of reasons, making the study of the process challenging. Two classes of event can signal a need for adaptation: 1) Events caused by one's own actions and specifically FeedBack -FB- from those actions (e.g. the investigators adapt their strategy after an erroneous choice), and 2) Events not linked to our actions, specifically Action-InDependent Events -AiDE- (e.g. the investigators adapt their strategy after a change of rule). These two types of information - FB and AiDE - will frequently occur concurrently. A critical and difficult part of adapting appropriately involves resolving the difference between the two. So for example an incorrect FB can occur because the investigators made an error, or because something unexpected in the environment has changed -the rule switched, someone cheated, etc. The Investigators must work out which it is, as they will frequently require different behavioral adaptations. Their task is made even more complex by the fact that the dynamics of evidence accumulation after FB vs AiDE are very different. FB has a direct temporal and causal link to an executed action, which means that the investigators are certain to derive information about a given action from a given FB. In contrast, AiDE have no such contiguity and no initial relation to actions, which means that the investigators must accumulate evidence to identify the appropriate adaptation to an AiDE. So the crucial dilemma is this: after an unwanted outcome, should the investigators adapt as if they made an error and received a negative FB, or should they continue to accumulate evidence as if there has been an AiDE to which they need to know how to adapt. Animals are able to resolve this credit assignment problem, as evidenced by their ability to appropriately adapt their behavior. A breakdown of this ability to link unexpected events to their correct cause would seem to be at the source of impairments in a wide range of psychological and neurological disorders, from addiction and OCD to psychological symptoms in Parkinson's disease. Yet the neural basis of this process is currently unknown, and FB and AiDE processing have been assessed separately so far. ADAPCO will provide unprecedented characterization of brain systems critically involved in learning from and adapting to FB, AiDE, and their interactions, thanks to fMRI studies.

ELIGIBILITY:
Inclusion Criteria:

* being able to provide a written consent form
* having a social insurance
* have a normal vision (with or without corrections)
* Right-handed

Exclusion Criteria:

* Subjects with MRI contraindications (e.g. pacemaker, claustrophobia, metal in the body, etc…).
* Subjects must be willing to be advise in case of discovery of brain abnormality.
* History of neurological or psychiatric illness
* Pregnant or nursing women
* Persons under guardianship, curatorship or any other administrative or judicial measure of deprivation of liberty

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-09-24 (Actual); Primary Completion 2022-08-24 (Estimated); Study Completion 2022-09-24 (Estimated)

PRIMARY OUTCOMES:
Behavioral data | 3 years
  Performance in the task will be assessed. Only subjects with performance in the task >80% in the last functional run will be included in the final analysis.
fMRI data | 3 years
  BOLD signal will be analyzed in relation to the events of the task of all subjects. Images must be not too much distorted to allow data analysis. As such, if a subject moved too much (translation>10mm; rotation>5°) the corresponding data will be excluded from the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Domenech, MD, Principal Investigator — Henri Mondor University Hospital
Locations (1):
- Hôpital Henri Mondor, Créteil, France